CLINICAL TRIAL: NCT02367014
Title: Phase 1/2 Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending-Dose Clinical Study for the Safety, Tolerability, and Efficacy of IV MTP-131 for Mitochondrial Myopathy in Genetically Confirmed Mitochondrial Disease
Brief Title: Safety, Tolerability, and Efficacy of MTP-131 for the Treatment of Mitochondrial Myopathy
Acronym: MMPOWER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIMM-201
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Mitochondrial Myopathy
Keywords: Mitochondrial Myopathy; Primary Mitochondrial Disease; Bendavia™; elamipretide
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose (Experimental): elamipretide 0.01 mg/kg/hr infused for 2 hours for 5 days
  Interventions: Drug: elamipretide (low dose)
- Intermediate dose (Experimental): elamipretide 0.10 mg/kg/hr infused for 2 hours for 5 days
  Interventions: Drug: elamipretide (intermediate dose)
- High dose (Experimental): elamipretide 0.25 mg/kg/hr infused for 2 hours for 5 days
  Interventions: Drug: elamipretide (high dose)
- Placebo (Placebo Comparator): In each cohort, subjects received either IV elamipretide given once daily for 2 hours for 5 days or matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: elamipretide (low dose) — elamipretide (0.01 mg/kg/hr) administered as single day intravenous infusion over 2 hours for 5 days
  Other Names: MTP-131
  Arms: Low Dose
Drug: elamipretide (intermediate dose) — elamipretide (0.10 mg/kg/hr) administered as single day intravenous infusion over 2 hours for 5 days
  Other Names: MTP-131
  Arms: Intermediate dose
Drug: elamipretide (high dose) — elamipretide (0.25 mg/kg/hr) administered as single day intravenous infusion over 2 hours for 5 days
  Other Names: MTP-131
  Arms: High dose
Drug: Placebo — placebo (at each dose cohort) administered as single day intravenous infusion over 2 hours for 5 days
  Arms: Placebo

SUMMARY:
Phase 1/2, multi-center, randomized, double-blind, multiple ascending dose, placebo-controlled study that enrolled 36 subjects with mitochondrial myopathy associated with genetically confirmed mitochondrial disease to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of MTP-131 in this patient population.

DETAILED DESCRIPTION:
This multi-center, randomized, double-blind, placebo-controlled study enrolled 36 subjects into 3 cohorts of 12 subjects each to evaluate treatment with 3 ascending doses of intravenous elamipretide (0.01, 0.10, and 0.25 mg/kg/hr infused for 2 hours). After each cohort, a Safety Monitoring Board (SMB) determined if dose escalation to the next higher dose of elamipretide was warranted. Each cohort went through 3 distinct periods: Screening, Treatment, and Follow-up.

The Screening Period started with informed consent and may have lasted up to 40 days. During this period, screening procedures to determine subject eligibility for the study occurred, including confirmation of disease, which incorporated a committee review of the investigator-submitted diagnosis and genetic results. The Treatment Period began on Day 1 (Visit 2) and lasted for 5 days (until Day 5 [Visit 6]). Within each cohort, 9 subjects were randomized to active drug and 3 subjects were randomized to placebo on Day 1 and subjects received treatment once a day for 5 consecutive days. Safety, tolerability, and efficacy measures were performed at pre-specified times. The Follow-up Period began at the time of discharge on Day 5. Subjects returned to the study center for the Follow-up Visit on Day 7 (+1 day).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mitochondrial disease believed to impair the mitochondrial respiratory chain.
* Eligibility requires prior genetic confirmation of mitochondrial disease.
* Diagnosis of mitochondrial myopathy judged by the Investigators to be due to existing mitochondrial disease.
* Must be able to complete a Screening Visit 6MWT.
* Body mass index (BMI) score >15.0 and <35.0 kg/m2 at Screening Visit.
* Women of childbearing potential must agree to use birth control as specified in the protocol from the date they sign the ICF until two months after the last dose of study drug.

Exclusion Criteria:

* Any prior or current medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements.
* Had any exclusionary Newcastle Mitochondrial Disease Adult Scale (NMDAS) scores at Screening Visit.
* Hospitalized (admitted as in-patient) within 1 month prior to the Baseline Visit.
* A history of type 1 diabetes mellitus (T1DM).
* Uncontrolled Type 1 (T1DM) or Type 2 diabetes mellitus (T2DM), in the opinion of the investigator.
* A creatinine clearance <45 mL/min as calculated by the Cockcroft Gault equation.
* Requires pacemaker, defibrillator, or has undergone cardiac surgery within 2 years of Screening Visit.
* QTc elongation defined as a QTc >450 msec in male subjects and >480 msec in female subjects.
* Uncontrolled hypertension (>160 mmHg systolic or >100 mmHg diastolic) at Screening Visit.
* History of rhabdomyolysis defined as an acute rise in the serum creatine phosphokinase (CPK) value that, in the opinion of the investigator, caused clinically significant symptoms.
* Serum sodium more than 5 meq/L below the reference lower limit of normal at Screening Visit.
* Participated in another interventional clinical trial within 3 months of the screening visit or is currently enrolled in a non-interventional clinical trial judged by the Investigator to be incompatible with the current trial.

  * Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Pittsburg of UPMC, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Centers: Akron Children's Hospital; Massachusetts General Hospital; University of Pittsburgh School of Medicine; University of California, San Diego
Groups:
- Low Dose: MTP-131: MTP-131 (low dose) 0.01 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- Intermediate Dose: MTP-131: MTP-131 (intermediate dose) 0.10 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- High Dose: MTP-131: MTP-131 (high dose) 0.25 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- Placebo: Placebo: Placebo Comparator (at each dose cohort) administered as single day intravenous infusion over 2 hours for 5 days
Period: Overall Study
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose: MTP-131: MTP-131 (low dose) administered as single day intravenous infusion over 2 hours for 5 days
- Intermediate Dose: MTP-131: MTP-131 (intermediate dose) administered as single day intravenous infusion over 2 hours for 5 days
- High Dose: MTP-131: MTP-131 (high dose) administered as single day intravenous infusion over 2 hours for 5 days
- Total: Total of all reporting groups
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.32) | 45.0 (14.09) | 42.3 (16.84) | 41.9 (15.83) | 42.5 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 6 | 9 | 30
  Male | 2 | 1 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Distance Walked (Meters) on the 6-minute Walk Test (6MWT)
Description: Change in distance walked as measured by meters on the 6-minute walk test from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Assessed at Baseline, Day 5 (end-of-treatment visit)
Measure: Least Squares Mean (Full Range); unit: meters
Groups:
- Low Dose: MTP-131 (low dose) 0.01 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- Intermediate Dose: MTP-131 (intermediate dose) 0.10 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- High Dose: MTP-131 (high dose) 0.25 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- Placebo: Placebo Comparator (at each dose cohort) administered as single day intravenous infusion over 2 hours for 5 days
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
meters | 13.5 [-72 to 86] | 36.5 [-20 to 107] | 64.5 [4 to 133] | 20.4 [-37 to 90]

2. Secondary Outcome: Change in Maximum Oxygen Uptake (ml/kg/Min)
Description: Change in maximum oxygen uptake as measured by mL/kg/min from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: All participants for whom maximum oxygen uptake was measured at baseline and Day 5
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- Intermediate: MTP-131 (intermediate dose) 0.10 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
- High: MTP-131 (high dose) 0.25 mg/kg/hour administered as single day intravenous infusion over 2 hours for 5 days
Arm/Group | Low Dose | Intermediate | High | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 6
ml/kg/min | 0.35 (2.617) | 2.36 (2.714) | 0.64 (3.121) | 2.14 (3.137)

3. Secondary Outcome: Change in Ventilatory Efficiency (VE/VCO2 Slope)
Description: Change in ventilatory efficiency as measured by the VE/VCO2 slope from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: All participants for whom VE/VCO2 slope measurements were recorded at Baseline and Day 5
Measure: Mean (Standard Deviation); unit: VE/VCO2 slope
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 6
VE/VCO2 slope | 0.749 (2.9412) | -0.671 (5.4024) | -1.681 (3.2834) | -1.375 (5.5801)

4. Secondary Outcome: Change in Aerobic Efficiency (ΔO2 Consumption/Δ Work Ratio)
Description: Change in aerobic efficiency as measured by ΔO2 consumption/Δ work ratio from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: All participants for whom aerobic efficiency measurements were recorded at Baseline and Day 5
Measure: Mean (Standard Deviation); unit: ΔO2 consumption/Δwork ratio
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 7 | 6
ΔO2 consumption/Δwork ratio | -0.234 (4.3414) | 0.643 (2.7507) | -0.214 (1.9727) | 0.738 (3.5959)

5. Secondary Outcome: Change in Oxygen Utilization (ΔVO2/ΔlogVE Ratio)
Description: Change in oxygen utilization as measured by ΔVO2/ΔlogVE ratio from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: All participants for whom oxygen utilization measurements were recorded at Baseline and Day 5
Measure: Mean (Standard Deviation); unit: ΔVO2/ΔlogVE ratio
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 7 | 7 | 8 | 6
ΔVO2/ΔlogVE ratio | -118.87 (229.105) | 184.99 (410.093) | 90.13 (116.281) | 166.50 (479.145)

6. Secondary Outcome: Change in Oxygen Uptake Kinetics (Mean Response Time as Measured by Seconds)
Description: Change in oxygen uptake kinetics (mean response time) as measured by seconds from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom oxygen uptake kinetics was measured
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Low Dose | Intermediate | High | Placebo
Number analyzed (Participants) | 7 | 7 | 8 | 6
seconds | 6.40 (11.402) | -2.49 (26.830) | -9.75 (26.288) | -7.47 (14.357)

7. Secondary Outcome: Change in Pre-exercise Lactate Levels (mg/dL)
Description: Change in pre-exercise lactate levels as measured by mg/dL from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom pre-exercise lactate levels were measured
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 6 | 8 | 6
mg/dL | 3.4 (9.00) | 13.8 (18.30) | 0.4 (10.25) | 4.4 (14.06)

8. Secondary Outcome: Change in Post-exercise Lactate Levels (mg/dL)
Description: Change in post-exercise lactate levels as measured by mg/dL from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom post- exercise lactate levels were measured
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 6 | 8 | 7
mg/dL | 6.9 (11.87) | 10.6 (42.93) | 4.3 (22.10) | 8.4 (13.21)

9. Secondary Outcome: Change in Peak Respiratory Exchange Ratio (VCO2/VO2)
Description: Change in peak respiratory exchange ratio as measured by VCO2/VO2 from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak respiratory exchange ratio was measured.
Measure: Mean (Standard Deviation); unit: VCO2/VO2 ratio
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 6
VCO2/VO2 ratio | 0.109 (0.0741) | 0.114 (0.1803) | 0.010 (0.0561) | 0.133 (0.1297)

10. Secondary Outcome: Change in Peak Respiratory Rate (Breaths/Min)
Description: Change in peak respiratory rate as measured by breaths/min from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak respiratory rate was measured
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 6 | 8 | 5
breaths/min | 1.4 (6.54) | -0.7 (5.72) | 0.9 (6.24) | 8.2 (5.26)

11. Secondary Outcome: Change in Peak Ventilation (L/Min)
Description: Change in peak ventilation as measured by L/min from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak ventilation was measured.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 6
L/min | 2.70 (8.692) | 8.87 (7.975) | 2.49 (8.303) | 8.47 (8.564)

12. Secondary Outcome: Change in Peak Heart Rate (Beats/Min)
Description: Change in peak heart rate as measured by beats per minute from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak heart rate was measured
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 8
beats/min | 10.1 (11.15) | 16.7 (13.02) | 4.5 (9.58) | 3.8 (7.85)

13. Secondary Outcome: Change in Peak Oxygen Saturation (% O2-saturated Hemoglobin)
Description: Change in peak oxygen saturation as measured by percentage of O2-saturated hemoglobin from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak oxygen saturation was measured.
Measure: Mean (Standard Deviation); unit: percentage of O2-saturated hemoglobin
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 7
percentage of O2-saturated hemoglobin | 0.0 (1.69) | 0.1 (1.07) | 0.6 (0.74) | 0.3 (1.60)

14. Secondary Outcome: Change in Peak Systolic Blood Pressure (mmHg)
Description: Change in peak systolic blood pressure as measured by mmHg from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak systolic blood pressure was measured.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 7
mmHg | 16.7 (21.00) | -1.5 (36.47) | 16.0 (12.71) | -2.7 (21.84)

15. Secondary Outcome: Change in Peak Diastolic Blood Pressure (mmHg)
Description: Change in peak diastolic blood pressure as measured by mmHg from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak diastolic blood pressure was measured
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 7
mmHg | 0.6 (12.67) | -1.4 (11.13) | -2.5 (9.07) | -6.6 (12.74)

16. Secondary Outcome: Change in Peak Borg Dyspnea
Description: Change in peak Borg dyspnea as measured by 0-10 with 0 meaning no breathlessness and 10 meaning maximal breathlessness from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom peak Borg dyspnea was measured.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 7
Units on a scale | -2.00 (2.00) | -2.2 (2.23) | -1.4 (1.30) | -0.4 (1.70)

17. Secondary Outcome: Change in VO2 Anaerobic Threshold (mL)
Description: Change in VO2 anaerobic threshold as measured by mL from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom VO2 was measured.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 5 | 7 | 4
mL | 30.00 (83.93) | 10.8 (80.35) | 1.6 (42.17) | 42.0 (51.89)

18. Secondary Outcome: Change in Watts
Description: Change in watts from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom watts was measured
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 8 | 7 | 8 | 8
watts | 9.6 (14.15) | 13.9 (12.48) | 5.4 (10.03) | 4.4 (11.87)

19. Secondary Outcome: Change in Temperature (°C)
Description: Change in temperature as measured by units of Celsius from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom temperature was measured
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 9
°C | -0.3 (0.54) | 0.2 (0.42) | 0.1 (0.28) | 0.0 (0.67)

20. Secondary Outcome: Change in ECG-PR Interval (Msec)
Description: Change in PR interval as measured by ECG in milliseconds from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom PR interval was measured
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 8 | 9 | 9
msec | -3.2 (7.77) | 8.3 (7.05) | 9.1 (9.55) | -1.6 (15.61)

21. Secondary Outcome: Change in ECG-QRS Complex (Msec)
Description: Change in QRS complex as measured by ECG in msec from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom QRS complex was measured
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
msec | 1.2 (7.14) | 2.3 (6.56) | -2.2 (8.86) | 0.8 (5.78)

22. Secondary Outcome: Change in ECG-QT Interval (Msec)
Description: Change in QT interval as measured by ECG in msec from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom QT interval was measured
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
msec | -6.0 (30.53) | -4.8 (12.94) | -16.7 (81.02) | -1.3 (18.49)

23. Secondary Outcome: Change in ECG-QTc Interval (Msec)
Description: Change in QTc interval as measured by ECG in msec from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom QTc interval was measured
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
msec | 3.4 (20.17) | 1.3 (20.24) | -23.2 (77.53) | 6.7 (17.28)

24. Secondary Outcome: Number of Participants Who Had Suicide Ideation, Suicidal Behavior, or Non-suicidal Self-injurious Behavior Post-screening.
Description: Number of participants with suicide ideation, suicidal behavior, or non-suicidal self-injurious behavior post-screening as measured on Days 1-5, and Day 7 on the Columbia Suicide Severity Rating Scale (CSSRS). A yes/no binary response is utilized in the following ten categories: 1 - Wish to be Dead; 2 - Non-specific Active Suicidal Thoughts; 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan; 5 - Active Suicidal Ideation with Specific Plan and Intent; 6 - Preparatory Acts or Behavior; 7 - Aborted Attempt; 8 - Interrupted Attempt; Category 9 - Actual Attempt (non-fatal); 10 - Completed Suicide. A yes/no binary response is also utilized in assessing self-injurious behavior without suicidal intent. A lower score means a better outcome whereas a higher score means a worse outcome.
Time Frame: Days 1-5 and Day 7.
Population: Participants for whom CSSR was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

25. Secondary Outcome: Change in Creatine Phosphokinase (IU/L)
Description: Change in Creatine Phosphokinase as measured by IU/L from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom creatine phosphokinase was measured
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
IU/L | -24.8 (25.10) | -161.7 (176.49) | -101.2 (149.07) | -154.9 (232.99)

26. Secondary Outcome: Change in Alanine Aminotransferase (ALT) (U/L)
Description: Change in Alanine aminotransferase (ALT) as measured by (U/L) from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom Alanine aminotransferase was measured
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
U/L | 19.3 (42.24) | -3.0 (4.92) | -5.3 (3.28) | 1.1 (5.80)

27. Secondary Outcome: Change in Aspartate Aminotransferase (AST) (U/L)
Description: Change in aspartate aminotransferase (AST) as measured by U/L from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom aspartate aminotransferase was measured
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9
U/L | 5.6 (9.93) | -2.2 (10.38) | -12.6 (18.08) | -4.4 (13.07)

28. Secondary Outcome: Change in Eosinophils (10^9 Cells/L)
Description: Change in eosinophils as measured by (10^9 cells/L) from baseline (last assessment prior to start of study) to Day 5 (end of treatment visit).
Time Frame: Baseline, Day 5
Population: Participants for whom eosinophils was measured
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 9
10^9 cells/L | 0.06 (0.073) | 0.08 (0.097) | -0.01 (0.064) | 0.04 (0.088)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Low Dose | Intermediate Dose | High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 7/9 | 5/9 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose (N=9) | Intermediate Dose (N=9) | High Dose (N=9) | Placebo (N=9)
Headache (Nervous system disorders) | 1 | 1 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
CPET was not performed on all subjects.Sensitivity analysis on change from Baseline in pre-and post-exercise lactate levels was not completed.Data from study sites were combined for efficacy and safety analyses.No site- effect analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days